CLINICAL TRIAL: NCT00409721
Title: A Randomized, Double-blind, Dose Ranging Study to Determine the Effect of Memantine on Functional Outcomes and Motor Neuron Degeneration in Patients With ALS
Brief Title: The Effect of Memantine on Functional Outcomes and Motor Neuron Degeneration in Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: ALS Association (Other)
Responsible Party: Sanjay Kalra, MD, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1204; EB2006ALS
Record Dates: First submitted 2006-12-08; First posted 2006-12-11 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2011-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; ALS; Motor Neuron Disease; MND; Memantine
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Memantine Low Dose (Experimental)
  Interventions: Drug: Memantine
- Memantine High Dose (Experimental)
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine

SUMMARY:
The purpose of the study is to investigate the effects of memantine in ALS patients using functional outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* El Escorial Classification of laboratory supported probable, probable,or definite ALS
* Age 18 - 80 years,
* ALS symptoms for no more than 3 years,
* FVC greater than or equal to 60% predicted,
* Riluzole naïve or have been on a stable dose of Riluzole for at least 2 months,
* Patients must have the ability to attend monthly study visits in Edmonton or Calgary, Alberta

Exclusion Criteria:

* Presence of significant sensory abnormalities, dementia, other neurologic diseases, uncompensated medical illness and psychiatric illness
* Female patients who are breastfeeding
* Use of concurrent investigational drugs,
* Patient unlikely to comply with study requirements
* Poor adherence to study protocol during run-in phase

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2007-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
ALS Functional Rating Scale-Revised (ALSFRS-R)
Forced vital capacity (FVC)
Manual Muscle Testing (MMT)
Addenbrooke Cognitive Examination (ACE)

SECONDARY OUTCOMES:
Motor unit number estimates of hand and foot muscles
N-acetylaspartate in the motor cortex

CONTACTS AND LOCATIONS:
Overall Officials: Ming Chan, MD, Principal Investigator — University of Alberta; Sanjay Kalra, MD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - Calgary ALS Neuromuscular Clinic, Calgary, Alberta
  - University of Alberta ALS Clinic, Edmonton, Alberta

REFERENCES:
- See also: ALS Association of America (ALSA) — http://www.alsa.org
- See also: ALS Society of Alberta — http://www.alsab.ca/
- See also: ALS Society of Canada — http://www.als.ca/